CLINICAL TRIAL: NCT05072626
Title: Study on High Medium-chain Triglyceride Nutritional Support in Infants With Biliary Atresia After Kasai Portoenterostomy
Brief Title: High Medium-chain Triglyceride Nutritional Support in Infants With Biliary Atresia
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Qian Tian, Deputy Director of clinical Nutrition, Children's Hospital of Fudan University
Other Study IDs: （2020）287
Record Dates: First submitted 2021-09-13; First posted 2021-10-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Biliary Atresia; Infant; Nutrition Support; Medium-chain Triglyceride
Keywords: Biliary Atresia; Kasai portoenterostomy; Nutrition Support; medium-chain triglyceride
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- high MCT formula nutritional support: Infants aged 0-3 months who underwent Kasai operation for congenital biliary atresia and were able to receive enteral nutrition through oral or tube feeding were administered a high MCT formula powder + breast milk (with the high MCT formula powder accounting for ≥50%) after the Kasai operation. If breast milk was insufficient, regular formula was used as a substitute. The recommended energy intake was set at 100-130% of DRIs.

SUMMARY:
This study is a prospective, single center and observational open clinical study.

DETAILED DESCRIPTION:
Biliary atresia (BA) is a significant disease leading to liver failure in infancy, with BA accounting for 50% of infant liver transplantation cases. Many BA children experience complications related to malnutrition, particularly during the first year of life. These complications are primarily characterized by reduced muscle mass and structural protein, impaired bone mineralization, diminished fat reserves, and deficiencies in vitamins and trace elements. Some studies have indicated that oral administration of specialized medium-chain triglycerides (MCT) and branched-chain amino acids FSMP with polysaccharides still result in malnutrition and growth retardation among BA children, necessitating enteral nutrition support treatment through tube feeding. The American Association for the Study of Biliary Atresia conducted a study on the prognosis of 104 children with biliary atresia after Kasai surgery across six clinical centers. They found that the key period for changes in growth rate occurred six months post-surgery, with faster-growing children exhibiting better prognoses compared to those with slower growth rates. Active nutritional therapy can enhance the prognosis of children with biliary atresia, particularly before and after Kasai surgery within the initial six-month period following surgery. Currently, there is no standardized process for using Foods for Special Medical Purpose in China nor any regulations governing the addition and monitoring of trace elements and vitamins. Therefore, this study aims to improve overall outcomes for children with biliary atresia through standardized nutrition assessment procedures as well as education, intervention, and follow-up measures.A total of 300 hospitalized patients were enrolled, all of whom received high MCT formula nutritional support following the Kasai operation, in order to investigate the impact of high MCT formula on the nutritional status and growth of children with biliary atresia after undergoing the Kasai procedure.

ELIGIBILITY:
Inclusion Criteria:

The Kasai procedure for infants with biliary atresia under the age of 3 months.

Exclusion Criteria:

* Complicated with cirrhosis, hepatitis, or other hepatic disorders;
* Complicated with other systemic serious diseases (such as congenital multiple malformations, chromosome abnormalities)

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The Kasai procedure for infants with biliary atresia under the age of 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Z-scores of body weight | 3 months after Kasai portoenterostomy
  The patient will be weighed in the recumbent position on an electronic infant scale. Z-scores for weight for age (WAZ) were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.

SECONDARY OUTCOMES:
Z-scores of body length | 1 month after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Z-scores of body length | 3 months after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Z-scores of body length | 6 months after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Z-scores of body length | 1 year after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Z-scores of body weight | 1 month after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Z-scores of body weight | 6 months after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Z-scores of body weight | 1 year after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Z-scores of head circumference | 1 month after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Z-scores of head circumference | 3 months after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Z-scores of head circumference | 6 months after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Z-scores of head circumference | 1 year after Kasai portoenterostomy
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
level of vitamin A | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin A | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin A | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin A | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of 25（OH) D | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of 25（OH) D | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of 25（OH） D | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of 25（OH） D | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin E | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin E | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin E | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin E | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin K | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin K | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin K | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
level of vitamin K | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Aspartate aminotransferase | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Aspartate aminotransferase | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Aspartate aminotransferase | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Aspartate aminotransferase | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Alanine aminotransferase | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Alanine aminotransferase | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Alanine aminotransferase | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Alanine aminotransferase | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Total Bilirubin | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Total Bilirubin | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Total Bilirubin | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Total Bilirubin | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Direct Bilirubin | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Direct Bilirubin | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Direct Bilirubin | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Direct Bilirubin | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Gamma-glutamyl transferase | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Gamma-glutamyl transferase | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Gamma-glutamyl transferase | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Gamma-glutamyl transferase | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Total bile acid | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Total bile acid | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Total bile acid | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Total bile acid | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
White blood cell | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
White blood cell | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
White blood cell | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
White blood cell | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
lymphocyte | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
lymphocyte | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
lymphocyte | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
lymphocyte | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Neutrophil count | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Neutrophil count | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Neutrophil count | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Neutrophil count | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
International Normalized Ratio | 1 month after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
International Normalized Ratio | 3 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
International Normalized Ratio | 6 months after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
International Normalized Ratio | 1 year after Kasai portoenterostomy
  Blood biochemical data are from clinical database.
Incidence of postoperative cholangitis | 1 year after Kasai portoenterostomy
  Data from clinical database
Liver transplantation | 1 year after Kasai portoenterostomy
  Data from clinical database
MMP-7 | 1 months after Kasai portoenterostomy
  Data from clinical database
MMP-7 | 3 months after Kasai portoenterostomy
  Data from clinical database
MMP-7 | 6 months after Kasai portoenterostomy
  Data from clinical database
MMP-7 | 1 year after Kasai portoenterostomy
  Data from clinical database
Intestinal flora | 1 months after Kasai portoenterostomy
  Data from clinical database
Intestinal flora | 3 months after Kasai portoenterostomy
  Data from clinical database
Intestinal flora | 6 months after Kasai portoenterostomy
  Data from clinical database
Intestinal flora | 1 year after Kasai portoenterostomy
  Data from clinical database
bile acid spectrum | 1 months after Kasai portoenterostomy
  Data from clinical database
bile acid spectrum | 3 months after Kasai portoenterostomy
  Data from clinical database
bile acid spectrum | 6 months after Kasai portoenterostomy
  Data from clinical database
bile acid spectrum | 1 year after Kasai portoenterostomy
  Data from clinical database

CONTACTS AND LOCATIONS:
Overall Officials: Tian Qian, M.D. PhD, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China